CLINICAL TRIAL: NCT06656806
Title: A Double-Blind, Placebo-Controlled, Single Center Study to Evaluate the Efficacy and Safety of Inhaled NC-107 As Compared to Placebo After 4 Weeks of Treatment in Patients with Anxiety
Brief Title: Efficacy and Safety of Inhaled NC-107 As Compared to Placebo After 4 Weeks of Treatment in Patients with Anxiety
Acronym: CALM
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Trinity Hypertension & Metabolic Research Institute (Other)
Collaborators: Nutraceutical Corporation (Unknown)
Responsible Party: Principal Investigator, Henry Anthony Punzi, Medical Director, Trinity Hypertension & Metabolic Research Institute
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NC-65-002
Record Dates: First submitted 2024-09-18; First posted 2024-10-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-09

CONDITIONS: Generalized Anxiety Disorder
Keywords: Generalized anxiety disorder; CBD; Metered dose inhaler
MeSH Terms: conditions — Generalized Anxiety Disorder

STUDY DESIGN:
Intervention Model Description: Double blinded Parallel Study
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Determine the presence and concentration of CBD in Subject's plasma with inhaled CBD (Active Comparator): Determine the presence and concentration of CBD in the plasma of male and female subjects with generalized anxiety disorder treated with inhaled CBD
  Interventions: Drug: Determine the presence and concentration of CBD in subject's plasma with inhaled CBD
- Measure concentrations of CBD is spot urine collections in subjects with inhaled CBD (Active Comparator): Measure concentration of CBD in spot urine collections in subject's with generalized anxiety disorder treated with inhaled CBD
  Interventions: Drug: Measure concentrations of CBD in spot urine collections from subjects treated with inhaled CBD

INTERVENTIONS:
Drug: Measure concentrations of CBD in spot urine collections from subjects treated with inhaled CBD — Measure concentrations of CBD in spot urine collections from subjects with generalized anxiety disorder treated with inhaled CBD
  Arms: Measure concentrations of CBD is spot urine collections in subjects with inhaled CBD
Drug: Determine the presence and concentration of CBD in subject's plasma with inhaled CBD — Determine the presence and concentration of CBD in plasma of subjects with generalized anxiety disorder treated with inhaled CBD
  Arms: Determine the presence and concentration of CBD in Subject's plasma with inhaled CBD

SUMMARY:
The goal of this clinical trial is to learn if inhaled drug NC-107 works to treat Generalized anxiety disorder in adults. It will also learn about the safety of the drug NC-107. The main questions it aims to answer are:

Does the inhaled drug NC-107 decrease the severity of anxiety in participants? What medical problems could participants have when taking drug NC-107? How quickly does NC-107 absorb and get into the blood stream? Researchers will compare drug NC-107 to a placebo (a look-alike substance that contains no drug) to see how effective NC-107 in treating generalized anxiety disorder.

Participants will be equal to or above 18 years of age and sign an informed consent. They will answer two questionnaires about anxiety and have vitals taken, as well as blood drawn for laboratory results. If a questionnaire reveals moderate anxiety and all blood work is normal the patient will enter the study. The patient will be instructed on the use of an inhaler, that will deliver the medication via the lung. Two puffs twice daily of NC-107 or placebo will be used during the remainder of the study.

Blood will be drawn for peak and trough levels of NC-107. Questionnaires will be completed at each visit.

ELIGIBILITY:
Inclusion Criteria

Inclusion Criteria:

Subjects must satisfy all the following criteria to be included in the study

1. Capable of reading, comprehending the consent process and providing written informed consent to participate in the study.
2. Male or female ≥ 18 years of age with generalized anxiety disorder. This includes a STAI ≥16 (moderate anxiety) or a GAD-7 score ≥10 (moderate anxiety).
3. Stable pharmacotherapeutics regimen with no change in the past 3 months.
4. Cannabis Naïve or abstinent from regular use (defined as >1x/month) for more than 6 months prior to the baseline visit.
5. Negative urine screen for metabolites of THC.
6. Women may be enrolled if all three of the following criteria are met:

   * Have a negative urine pregnancy test at screening, for females of childbearing potential.
   * Are not breastfeeding
   * Do not plan to become pregnant during the study And if one of the following three criteria is met
   * Have had a hysterectomy or tubal ligation at least 6 months prior to signing the informed consent form
   * Have been postmenopausal for at least 1 year
   * Are of childbearing potential and will practice one of the following methods of birth control throughout the study: oral, patch, injectable, or implantable hormone contraception, intrauterine device, diaphragm plus spermicide or female condom plus spermicide.

Exclusion Criteria:

1. Patients with severe hypertension (mean seated cuff diastolic blood pressure >115 mmHg or mean seated systolic blood pressure >180mmHg) or any form of secondary hypertension at time of screening
2. Patients within the past 6 months with a history of hypertensive encephalopathy, stroke, or transient ischemic attack.
3. Patients within the last 6 months with a history of myocardial infarction, percutaneous transluminal coronary revascularization, coronary bypass graft, valvular surgery or unstable angina.
4. Patients with a history of heart block greater than First Degree Sinoatrial Block. Wolff-Parkinson-White Syndrome, Sick Sinus Syndrome, Atrial Fibrillation, Atrial Flutter, Congestive Heart Failure, or other manifestations of clinically significant cardiac valvular disease.
5. Patients with hemo-dynamically significant cardiac valvular disease.
6. Patients with evidence of significant chronic renal impairment as indicated by a serum creatinine of > 2.5mg/dL at Screening.
7. Patients with evidence of liver disease as indicated by AST (SGOT) or ALT (SGPT) > 2.5 times or total bilirubin > 1.5 times, the upper limit of the laboratory normal range at Screening.
8. Patients who demonstrate other laboratory test values deviating from the normal range which are considered clinically significant by the investigator.
9. Patients with insulin and non-insulin dependent diabetes mellitus not controlled on diet, insulin or oral hypoglycemics as defined by a HgA1c >10.5 mg/dcL at Visit 1
10. Severe psychological or emotional condition ( Current substance abuse, major depressive, psychotic, and bipolar disorder) that are not associated with Generalized Anxiety Disorder which may interfere with participation in the study.
11. History of or current use of illicit drugs or alcohol abuse.
12. Participation in a clinical trial and taking any investigational drug within 30 days prior to enrolling into the study (Screening).
13. Any other medical condition which, in the Investigator's opinion, may render the patient unable to complete the study or which would interfere with optimal participation in the study or produce significant risk to the patient

    -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Measure the concentration of CBD in the plasma of subjects | 4 weeks
  Measure the concentration of CBD in the plasma of male and female subjects with Generalized Anxiety Disorder treated with inhaled CBD.

SECONDARY OUTCOMES:
Concentrations of CBD in spot urine collections. | 4 weeks
  Measure concentrations of CBD in spot urine collections from male and female subjects with Generalized Anxiety Disorder treated with inhaled CBD.

OTHER OUTCOMES:
Decrease in the levels of Anxiety with Questionnaires | 4 weeks
  Whether there is a decrease in the levels of anxiety in the STAI and or GAD-7 questionnaires at weeks 1, 2, 3, and 4, when compared to baseline week 0.

CONTACTS AND LOCATIONS:
Locations (1):
- Punzi Medical Center, Carrollton, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Phase 1 clinical trial